CLINICAL TRIAL: NCT02811341
Title: A Clinical Analysis of Scopolamine Hydrobromide in Probe-based Confocal Laser Endomicroscopy for Gastroendoscopy Examination
Brief Title: The Application of Spasmolytic in PCLE Examination of Superior Gastrointestinal Endoscope
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2015SDU-QILU-G01
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Using Copolamine Butylbromide in Probe-based Confocal Laser Endomicroscopy for Gastroendoscopy Examination
Keywords: Scopolamine butylbromide PCLE
MeSH Terms: interventions — Scopolamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A group (Placebo Comparator): Using normal saline before pcle examination
  Interventions: Drug: normal saline
- B group (Experimental): Using Scopolamine Hydrobromide before pcle examination
  Interventions: Drug: Scopolamine Hydrobromide

INTERVENTIONS:
Drug: Scopolamine Hydrobromide
  Arms: B group
Drug: normal saline
  Arms: A group

SUMMARY:
Scopolamine butylbromide might be helpful for the outcome of superior gastrointestinal endoscope examination.

DETAILED DESCRIPTION:
The peristalsis of gastrointestinal tract has a adverse affection on the process of the PCLE examination .Scopolamine butylbromide is a widely used spasmolytic，which can reduce the peristalsis of gastrointestinal tract effectly.The application of it may benefit the images'quality ,the acurrate of diagnosis and shorten the examination time.

ELIGIBILITY:
Inclusion Criteria:

* outpatients attending endomicroscopy
* able to give written informed consent

Exclusion Criteria:

* coagulopathy
* acute upper digestive tract bleeding
* pregnancy or breast feeding
* allergy to fluorescein sodium
* impaired renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
endomicroscopic image quality | 7months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD.PhD., Principal Investigator — Qilu Hospital of Shandong University; Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No